CLINICAL TRIAL: NCT04186949
Title: Early Origins of Allergy and Asthma
Acronym: ARIES
Status: Completed | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Chile (Other); Comisión Nacional de Investigación Científica y Tecnológica (Other Government)
Responsible Party: Sponsor
Other Study IDs: ACT172097; 170925013 (Other: Comité Ético Científico, Pontificia Universidad Católica de Chile)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-03

CONDITIONS: Allergy; Asthma; Food Allergy; Allergic Sensitisation; Atopic Dermatitis
Keywords: birth cohort; Chile
MeSH Terms: conditions — Hypersensitivity; Asthma; Food Hypersensitivity; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Birth cohort study with recruitment during pregnancy to determine prenatal and perinatal conditions, as well as genetic and epigenetic factors, that participate in the early setting of immune responses, and the role of these in the later determination of the risk of allergic diseases, asthma, and metabolic conditions in the offspring.

DETAILED DESCRIPTION:
Despite recent advances in the understanding of the pathogenesis of allergies and asthma, these diseases still have no clear preventative measures or curative treatments. Growing evidence shows that atopic dermatitis (AD), food allergy (FA), allergic rhinitis, and asthma are largely determined during the first 1000 days (time elapsed from conception to the 2nd birthday). This cohort aims to determine prenatal and perinatal conditions, as well as genetic and epigenetic factors, that participate in the early setting of immune responses, and the role of these in the later determination of the risk of allergic diseases, and asthma in the offspring.

The investigators have designed a birth cohort of 250 families with recruitment in pregnancy (~14 weeks). The plan is to genotype relevant allergy/asthma-associated variants and will perform immunophenotyping and evaluation of allergy biomarkers in cord blood. At 2 years of age the investigators will assess if infants have developed allergic sensitization, AD, FA, as well as biomarkers of asthma including the asthma predictive index. The study will also evaluate how maternal conditions modify immune programming through epigenetic modifications, and will then confirm newborn epigenetic cues of allergy/asthma risk. Next, the investigators will assess composition/diversity of maternal gut, placenta, breastmilk and infant gut microbiome and their association with immunophenotype and biomarkers at birth, and clinical outcomes at age 2. Finally, another specific objective is to assess how environmental exposures (perinatal outdoor and indoor pollution, endotoxin and allergens) affect the incidence of allergic sensitization, AD, FA, and risk of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women living in Chile's central regions
* Offspring of women recruited in the cohort study

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women living in Chile's central regions (i.e. mothers), their partners (i.e. fathers), and their offspring.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Development of allergic diseases in offspring | 2 years
  Atopic dermatitis, food allergy, allergic sensitization, predicted increased risk of asthma

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Borzutzky, M.D., Study Director — Pontificia Universidad Catolica de Chile; Paul Harris, M.D., Principal Investigator — Pontificia Universidad Catolica de Chile; Paola Casanello, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile; José A Castro-Rodriguez, M.D. PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez CD, Casanello P, Harris PR, Castro-Rodriguez JA, Iturriaga C, Perez-Mateluna G, Farias M, Urzua M, Hernandez C, Serrano C, Sandoval M, Hoyos-Bachiloglu R, Uauy R, Borzutzky A. Early origins of allergy and asthma (ARIES): study protocol for a prospective prenatal birth cohort in Chile. BMC Pediatr. 2020 Apr 15;20(1):164. doi: 10.1186/s12887-020-02077-x. PMID 32293348